CLINICAL TRIAL: NCT06048315
Title: A Single Center, Single Arm Clinical Study on the Treatment of Advanced Non-small Cell
Brief Title: A Single Center, Single Arm Clinical Study on the Treatment of Advanced Non-small Cell Lung Cancer With Positive EGFR Sensitive Mutations and Failed EGFR TKIs With the Combination of Enrotinib and Paclitaxel Monoclonal Antibody
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Degan Lu (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor-Investigator, Degan Lu, chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2023(091)
Record Dates: First submitted 2023-09-10; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer; TKI Resistance; EGFR Sensitive Mutation; Anlotinib; Pianzumab
MeSH Terms: conditions — Lung Neoplasms | interventions — anlotinib; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Anlotinib — Every 3 weeks is a treatment cycle, starting from the first day of each treatment cycle with oral administration of 12mg of arotinib once a day, stopping for one week after taking it for two weeks until disease progression (PD), unacceptable toxic reactions, withdrawal of informed consent, end of study, loss of follow-up or death, whichever occurs first.
  Other Names: Frikovi
Drug: Penpulimab — On the first day, Pianzumab (200mg intravenous infusion) was administered every 3 weeks until disease progression (PD), unacceptable toxic reactions, withdrawal of informed consent, end of study, loss of follow-up or death, whichever occurs first.
  Other Names: Anico

SUMMARY:
Lung cancer is the second most common malignancy and mortality rate in the world. In the United States and Europe, approximately 10% to 15% of NSCLC patients have epidermal growth factor receptor (EGFR)-sensitive mutations, with higher mutation rates of 30% to 40% in Asia, and objective response rates (ORRs) of 76% to 80% with EGFR Tyrosine Kinase Inhibitor (TKI)-targeted therapy. However, resistance mechanisms such as EGFR, MET, PIK3CA and BRAF gene alterations occur with the development of resistance to EGFR-TKI therapy; Median Progression Free Survival (mPFS) for only 2.8-3.2 months; The median overall survival (mOS) is only 7.5-10.6 months. Due to the variety of mechanisms of resistance to EGFR-TKIs and the limited efficacy of chemotherapy, it is necessary to provide salvage treatment for advanced non-small cell lung cancer that is positive for EGFR-sensitive mutations and has failed EGFR TKIs.

Anlotinib is a novel multi-target tyrosine kinase inhibitor (TKI) used to inhibit tumor angiogenesis and proliferative signaling. The main targets of anlotinib include tyrosine kinase vascular endothelial growth factor receptor 1-3 (VEGFr1-3), fibroblast growth factor receptor 1-4 (Fibroblast Growth Factor Receptor 1-4), platelet-β derived growth factor receptor α and β, and stem cell factor receptor. Anlotinib is rapidly absorbed through the intestine, has high bioavailability, a half-life of 5 days, and is convenient for oral administration, which is conducive to improving patient dependence. IN MAY 2018, THE CHINA FOOD AND DRUG ADMINISTRATION APPROVED ANLOTINIB FOR MARKETING, ENTERED THE MEDICAL INSURANCE CATALOG IN OCTOBER OF THE SAME YEAR, AND WAS RECOMMENDED BY THE CHINESE SOCIETY OF CLINICAL ONCOLOGY (CSCO) FOR THE THIRD-LINE TREATMENT OF LUNG CANCER IN 2019.

Penpulimab is a humanized immunoglobulin G1 monoclonal antibody (IgG1), which is a class 1 new drug jointly developed by Zhongshan Akeso Biopharmaceutical Co., Ltd. and Chia Tai Tianqing Pharmaceutical Group Co., Ltd., which can specifically bind to PD-1 molecules on the surface of T lymphocytes, thereby blocking the PD-1/PD-L1 pathway that leads to tumor immune tolerance, and reactivating the anti-tumor activity of T lymphocytes to achieve the purpose of treating tumors. A number of preclinical in vitro trials have verified the effect of PEAMPLIMAB in blocking PD-1 pathway, and the results of preclinical pharmacodynamics, animal pharmacokinetics and toxicology have shown that PEAMPLIMAB has good stability, reduced host cell protein residues, and can effectively bind to antigens, and eliminate Fc-mediated effector function, with higher safety.

AK105-201 is a multicenter, double-blind, randomized controlled, phase III clinical trial evaluating the efficacy and safety of pianpulimab combined with carboplatin + paclitaxel in the first-line treatment of locally advanced or metastatic squamous non-small cell lung cancer, the primary endpoint of the study was PFS, and the secondary endpoint was OS, and the results showed that the mPFS group of pianpulimab and the control group were 7.6m and 4.2m, respectively, and the HR was 0.44, reducing the risk of disease progression by 56%. In the 2022 CSCO guidelines for the diagnosis and treatment of non-small cell lung cancer, peamplimab combined with platinum-containing chemotherapy is recommended as the first-line treatment for stage IV driver-free squamous cell carcinoma Grade II. In advanced patients with EGFR TKIs resistance, pemetrexed chemotherapy has a good efficacy, with a median PFS of 2.83 months and a response rate of 22%. The AK105-203 study is a multicenter phase II clinical study led by Professors Jiao Shun and Bai Li of the Chinese PLA General Hospital of the People's Liberation Army of Anlotinib combined with péamplimab in the first-line treatment of hepatocellular carcinoma, with a median follow-up of 23 months and mPFS of 8.8 months.

Therefore, based on the results of the current study on immunosuppressants and antiangiogenic drugs for the treatment of NSCLC, and the current research status in patients with advanced NSCLC who are positive for EGFR-sensitive mutations and have failed EGFR TKIs, we expect to conduct an exploratory clinical study of PD-1 antibody (péamplimab) combined with anlotinib in patients with advanced NSCLC who are positive for EGFR-sensitive mutations and have failed EGFR TKIs, with the aim of evaluating the safety of this combination, It was further investigated whether this combination could further improve the survival benefit of patients with advanced NSCLC.

DETAILED DESCRIPTION:
Non-small cell lung cancer is the most common type of lung cancer, accounting for 80%-85% of all lung cancers, and about 57% of patients with advanced NSCLC have distant metastases at the time of diagnosis, although chemotherapy, targeted therapy and anti-angiogenic drugs have become the cornerstone of the treatment of advanced NSCLC, but the emergence of immune checkpoint inhibitors in recent years has changed the treatment model of NSCLC. Immune checkpoint inhibitors enhance the body's antitumor activity by inhibiting the immune escape mechanism of tumors, and prolong the survival time of NSCLC patients. According to statistics, the 5-year survival rate of NSCLC patients who join immunotherapy and undergo multi-line therapy can reach 16%.

Previous studies have confirmed that anti-angiogenic drugs and immunotherapy have the effect of improving tumor microenvironment, basic translational and clinical studies have shown that immune checkpoint inhibitors and anti-angiogenic drugs have a synergistic effect, anti-angiogenic drugs can exert immunosuppressive effects by preventing immune invasion of tumors through tissue remodeling and fibrosis, and patients can benefit from PD-1/PD-L1 inhibitors combined with anti-angiogenic therapy.

In the CheckMate 057 and KEYNOTE-001 studies, the ORRs of patients with advanced NSCLC treated with anti-PD-1 monotherapy were 19% (mPFS 2.3 months) and 19.4% (mFS 3.7 months), respectively. The results of Wangpl et al. demonstrated that anti-PD-1 combined with anlotinib in the treatment of advanced NSCLC had an ORR of 28.4%, a DCR of 86.6%, and an mPFS of 6.9 months (95% CI, 5.5-8.3 months), confirming that the combination therapy of anlotinib and anti-PD-1 drugs has a good efficacy and can be used as a second- or third-line treatment in previously treated patients with advanced NSCLC, indicating VEGF-VEGFR2 and PD-1-/ The dual inhibition of the PD-L1 pathway has clinical applicability.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in clinical research, aged 18-75 years old, regardless of gender, and sign a written informed consent form.
* According to the International Association for the Study of Lung Cancer and the Joint Committee on the American Classification of Cancer, 8th edition TNM staging of lung cancer, locally advanced or metastatic (IIIB, IIIC, IV) NSCLC patients who are confirmed by histology or cytology to be inoperable and unable to undergo radical synchronous radiotherapy and chemotherapy.
* NSCLC patients who have tested positive for EGFR gene sensitive mutations through driver gene testing and have not undergone systematic treatment after EGFR TKI treatment failure.
* Newly treated patients who have not received systemic radiotherapy and chemotherapy in the past, or patients who have relapsed after more than 6 months of follow-up after adjuvant chemotherapy after surgery.
* At least one evaluable lesion judged according to RECIST criteria.
* Men or women aged 18 years ≤ 75 years old.
* ECOG PS 0 or 1.
* The expected survival period is ≥ 12 weeks.
* Adequate blood function: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L and platelet count ≥ 90 × 109/L and hemoglobin ≥ 9 g/dL.
* Adequate liver function: Serum bilirubin ≤ 1.5 times the upper limit of normal value (ULN); AST and ALT ≤ 2.5 times the upper limit of normal value (ULN); Alkaline phosphatase ≤ 5 times the upper limit of normal value (ULN).
* Adequate renal function: serum creatinine ≤ upper limit of normal (ULN) or calculated creatinine clearance rate ≥ 60 mL/min.
* Women of childbearing age must have negative pregnancy test results within 28 days prior to enrollment in the study (unless amenorrhea has occurred for 24 months). If the pregnancy test is more than 7 days after the first administration, a urine pregnancy test is required for validation (within 7 days before the first administration).
* If there is a risk of conception, all patients (whether male or female) are required to use contraceptive measures with an annual failure rate of less than 1% throughout the entire treatment period until 120 days after the last study drug administration.

Exclusion Criteria:

* Known hypersensitivity to any component contained in the formulation of arotinib or piazepril monoclonal antibody;
* Individuals who are intolerant to the treatment of investigational drugs or are known to be allergic to any investigational drug or its excipients.
* Pregnant or lactating women, or female patients with fertility who have not taken contraceptive measures;
* Existing severe acute infections that have not been controlled; Those who may have purulent or chronic infections, and the wound persists without healing;
* Individuals with previously severe heart disease, including congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina, myocardial infarction, severe heart valve disease, and refractory hypertension;
* Those who suffer from uncontrollable neurological, mental disorders or mental disorders, have poor compliance, and are unable to cooperate and describe treatment responses; Patients with primary brain tumors or central nervous system metastases whose condition has not been controlled and who have obvious intracranial hypertension or neuropsychiatric symptoms;
* Have coagulation dysfunction or bleeding tendency, or have a history of thrombotic or hemorrhagic diseases;
* Those undergoing anticoagulation or thrombolysis treatment;
* There are unhealed wounds, ulcers, or fractures;
* Currently participating in interventional clinical research treatment, or receiving other research drugs or using research instruments within 4 weeks before the first administration;
* Has undergone major surgical treatment (excluding surgery for biopsy purposes) within 4 weeks prior to the first study drug administration, or is expected to undergo major surgery during the study period;
* Pulmonary interstitial fibrosis with respiratory failure;
* Patients with chronic obstructive pulmonary disease and respiratory failure;
* Based on chest imaging examination, sputum examination, and clinical examination, it is determined that there is active pulmonary tuberculosis (TB) infection;
* Patients with active, known or suspected autoimmune diseases. Patients with hypothyroidism who only require hormone replacement therapy can be selected;
* Patients who require systemic corticosteroids (with a dose equivalent to>10 mg prednisone/day) or other immunosuppressive drugs within the 14 days prior to enrollment. Patients who use inhaled or topical corticosteroids, as well as patients with adrenal corticosteroid replacement therapy doses equivalent to>10 mg prednisone/day, may participate in the study if there is no active autoimmune disease;
* Previously received PD-1 or PD-L1 antibody treatment for any reason;
* Suffering from other primary malignant tumors before the start of the study;
* Other situations where the researcher believes that patients are not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | 12month
  It refers to the time from the patient signing the informed consent form to the earliest occurrence of tumor progression, including death from any cause.

SECONDARY OUTCOMES:
Overall Survival | 12month
  It refers to the time from the patient signing the informed consent form for participating in the study to the time of death due to any reason.
Objective Response Rate | 12month
  Refers to the proportion of patients with partial and complete remission in all patients.
Disease Control Rate | 12month
  The proportion of patients with partial, complete, and stable efficacy among all patients.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Zappa C, Mousa SA. Non-small cell lung cancer: current treatment and future advances. Transl Lung Cancer Res. 2016 Jun;5(3):288-300. doi: 10.21037/tlcr.2016.06.07. PMID 27413711
- [Result] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Result] Yang CJ, Hung JY, Tsai MJ, Wu KL, Liu TC, Chou SH, Lee JY, Hsu JS, Huang MS, Chong IW. The salvage therapy in lung adenocarcinoma initially harbored susceptible EGFR mutation and acquired resistance occurred to the first-line gefitinib and second-line cytotoxic chemotherapy. BMC Pharmacol Toxicol. 2017 May 10;18(1):21. doi: 10.1186/s40360-017-0130-0. PMID 28486985
- [Result] Han B, Li K, Zhao Y, Li B, Cheng Y, Zhou J, Lu Y, Shi Y, Wang Z, Jiang L, Luo Y, Zhang Y, Huang C, Li Q, Wu G. Anlotinib as a third-line therapy in patients with refractory advanced non-small-cell lung cancer: a multicentre, randomised phase II trial (ALTER0302). Br J Cancer. 2018 Mar 6;118(5):654-661. doi: 10.1038/bjc.2017.478. Epub 2018 Feb 13. PMID 29438373
- [Result] Errors in Number at Risk and Author Email Address. JAMA Oncol. 2018 Nov 1;4(11):1625. doi: 10.1001/jamaoncol.2018.5345. No abstract available. PMID 30419091
- [Result] Song Y, Zhou K, Jin C, Qian Z, Hou M, Fan L, Li F, Ding K, Zhou H, Li X, Chen B, Sun X, Song X, Jiang M, Zhang Q, Liu L, Yu G, Hu Y, Zhao Z, Liu L, Xue H, Luo J, He B, Jin X, Zhao M, Li B, Xia Y, Zhu J. Penpulimab for Relapsed or Refractory Classical Hodgkin Lymphoma: A Multicenter, Single-Arm, Pivotal Phase I/II Trial (AK105-201). Front Oncol. 2022 Jul 7;12:925236. doi: 10.3389/fonc.2022.925236. eCollection 2022. PMID 35875118
- [Result] Wang P, Fang X, Yin T, Tian H, Yu J, Teng F. Efficacy and Safety of Anti-PD-1 Plus Anlotinib in Patients With Advanced Non-Small-Cell Lung Cancer After Previous Systemic Treatment Failure-A Retrospective Study. Front Oncol. 2021 Mar 15;11:628124. doi: 10.3389/fonc.2021.628124. eCollection 2021. PMID 33791214
- [Result] Han C, Ye S, Hu C, Shen L, Qin Q, Bai Y, Yang S, Bai C, Zang A, Jiao S, Bai L. Clinical Activity and Safety of Penpulimab (Anti-PD-1) With Anlotinib as First-Line Therapy for Unresectable Hepatocellular Carcinoma: An Open-Label, Multicenter, Phase Ib/II Trial (AK105-203). Front Oncol. 2021 Jul 13;11:684867. doi: 10.3389/fonc.2021.684867. eCollection 2021. PMID 34327136